CLINICAL TRIAL: NCT05025319
Title: Optimization of Bedside Chest X-rays Taken in the Intensive Care Unit by Using Current Software-based Techniques
Status: Active, not recruiting | Type: Observational
Sponsor: Joint Authority for Päijät-Häme Social and Health Care (Other)
Collaborators: Tampere University (Other)
Responsible Party: Principal Investigator, Marjo Soini, Chief Physicist, Joint Authority for Päijät-Häme Social and Health Care
Other Study IDs: R19100 (PHKS)
Record Dates: First submitted 2021-08-26; First posted 2021-08-27 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: X-Rays
Keywords: Imaging; Grid; X-ray; Image quality
MeSH Terms: interventions — X-Rays

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Taditional Grid: Patients imaged with traditional grid
  Interventions: Radiation: X-ray image
- Virtual Grid: Patients imaged with virtual grid
  Interventions: Radiation: X-ray image

INTERVENTIONS:
Radiation: X-ray image — Bedside x-ray at intensive unit.

SUMMARY:
This study investigates how to utilize an algorithm-based virtual grid in lung imaging in intensive care unit patients. The aim is to compare the radiation dose caused by imaging with a virtual grid and a traditional grid and relate this to the achieved image quality. The study aims to determine how the radiation dose can be lowered and still obtain the same diagnostic image quality as using a traditional scatter-limiting lattice.

ELIGIBILITY:
Inclusion Criteria:

* All patients in the intensive care unit with an imaging of the lung.

Exclusion Criteria:

* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intensive care patients
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Image quality | 2 years
  Compare the radiation dose caused by imaging with a virtual grid and a traditional grid and relate this to the achieved image qualit

CONTACTS AND LOCATIONS:
Locations (1):
- Joint Authority for Päijät-Häme Social and Health Care, Lahti, Finland

IPD SHARING:
Plan to Share IPD: Undecided